CLINICAL TRIAL: NCT07405879
Title: The Impact of Having a Tattoo on Fertility Treatment Outcome: A Prospective Randomized Controlled Trial
Brief Title: The Impact of Having a Tattoo on Fertility Treatment Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Michael Dahan, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2026-11525
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Infertility; Assisted Reproductive Technology Outcomes
Keywords: In vitro fertilization; Embryo transfer; Live birth; pregnancy; Assisted reproductive technology; Tattoos; Chronic inflammation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tattoo Group: Participants undergoing IVF with planned embryo transfer who have one or more tattoos at the time of embryo transfer.
- No Tattoo Group: Participants undergoing IVF with planned embryo transfer who do not have any tattoos at the time of embryo transfer.

SUMMARY:
Tattoos are increasingly common among women of reproductive age, yet their potential systemic inflammatory effects and impact on fertility treatment outcomes are unknown. This prospective observational cohort study aims to evaluate whether the presence, size, duration, and ink characteristics of tattoos are associated with pregnancy outcomes following embryo transfer in women undergoing in vitro fertilization (IVF).

DETAILED DESCRIPTION:
This is a single-center, prospective observational cohort study conducted at the McGill University Health Centre Reproductive Centre. Women undergoing IVF with planned fresh or frozen blastocyst embryo transfer will be enrolled and categorized based on tattoo presence and characteristics. Tattoo information will be collected using a standardized questionnaire and direct measurement. Participants will be followed for pregnancy and obstetric outcomes through medical chart review. The primary outcome is ongoing pregnancy rate following embryo transfer. Secondary outcomes include clinical pregnancy, biochemical pregnancy, miscarriage, ectopic pregnancy, and live birth.

ELIGIBILITY:
Inclusion Criteria:

Women aged 21-40 years Undergoing IVF with planned fresh or frozen blastocyst embryo transfer Availability of good-quality blastocyst embryos Willingness to provide informed consent

Exclusion Criteria:

Significant untreated uterine abnormalities

≥3 prior failed embryo transfers Hydrosalpinx in situ BMI >40 kg/m² Age >41 years at embryo creation Submucosal fibroids in situ Use of medications affecting implantation (e.g., chronic steroids, metformin)

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of women aged 21 to 40 years undergoing in vitro fertilization (IVF) with a planned fresh or frozen blastocyst embryo transfer at a single academic fertility center. Eligible participants must have at least one good-quality blastocyst available for transfer and provide informed consent. Participants are prospectively followed and categorized based on the presence or absence of tattoos at the time of embryo transfer. Pregnancy and obstetric outcomes are assessed through review of medical records over the study follow-up period.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2031-01-28 (Estimated); Study Completion 2031-01-28 (Estimated)

PRIMARY OUTCOMES:
Ongoing Pregnancy Rate | 12 weeks gestation
  Presence of fetal heartbeat on ultrasound at ≥12 weeks

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6-8 weeks of gestation
  presence of a gestational sac
Biochemical pregnancy | 4-5 weeks of gestation
  positive BHCG test
Miscarriage rate | before the 20th week of pregnancy
  The spontaneous loss of a fetus
Ectopic pregnancy rate | upto 10 weeks of gestation
  the frequency at which a fertilized egg implants outside the uterine cavity
Live birth rate | over 23 weeks of gestation
  the frequency of successful deliveries resulting in at least one live-born infant

CONTACTS AND LOCATIONS:
Overall Officials: michael haim dahan, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- MUHC Reproductive Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves sensitive reproductive health information, and participants did not provide consent for public data sharing. In addition, the study is a single-center observational cohort, and data are retained in coded form in accordance with institutional ethics approval and privacy regulations.

REFERENCES:
- [Background] Xie J, Yan L, Cheng Z, Qiang L, Yan J, Liu Y, Liang R, Zhang J, Li Z, Zhuang L, Hao C, Wang B, Lu Q. Potential effect of inflammation on the failure risk of in vitro fertilization and embryo transfer among infertile women. Hum Fertil (Camb). 2020 Sep;23(3):214-222. doi: 10.1080/14647273.2018.1543898. Epub 2018 Nov 27. PMID 30477363
- [Background] Mukherjee N, Sharma R, Modi D. Immune alterations in recurrent implantation failure. Am J Reprod Immunol. 2023 Feb;89(2):e13563. doi: 10.1111/aji.13563. Epub 2022 May 29. PMID 35587052
- [Background] Islam PS, Chang C, Selmi C, Generali E, Huntley A, Teuber SS, Gershwin ME. Medical Complications of Tattoos: A Comprehensive Review. Clin Rev Allergy Immunol. 2016 Apr;50(2):273-86. doi: 10.1007/s12016-016-8532-0. PMID 26940693